CLINICAL TRIAL: NCT00981643
Title: The Effects of Meditation on Pain, Fatigue and Physical Functioning in Patients With Multiple Sclerosis and Peripheral Neuropathy
Brief Title: Effects of Meditation on Multiple Sclerosis and Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CCF 08-950
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2011-09

CONDITIONS: Multiple Sclerosis; Peripheral Neuropathy
Keywords: Meditation; Multiple Sclerosis; Peripheral Neuropathy
MeSH Terms: conditions — Multiple Sclerosis; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Multiple Sclerosis, Meditation group (Experimental): Multiple Sclerosis, Meditation instruction and practice group
  Interventions: Behavioral: Meditation instruction and practice
- Multiple Sclerosis, Control group (No Intervention): Multiple Sclerosis, Control group
- Peripheral Neuropathy, Meditation group (Experimental): Peripheral Neuropathy, Meditation instruction and practice group
  Interventions: Behavioral: Meditation instruction and practice
- Peripheral Neuropathy, Control group (No Intervention): Peripheral Neuropathy, Control group

INTERVENTIONS:
Behavioral: Meditation instruction and practice — Meditation techniques introduced and practiced, in a group setting, once weekly for 8 weeks
  Arms: Multiple Sclerosis, Meditation group; Peripheral Neuropathy, Meditation group

SUMMARY:
This study will evaluate the effects of mindfulness and concentration meditation on pain, fatigue, and physical functioning in patients with either multiple sclerosis or peripheral neuropathy.

DETAILED DESCRIPTION:
We propose a prospective, randomized controlled study evaluating the effects of mindfulness meditation and concentration meditation on pain, fatigue, and physical functioning in patients with either multiple sclerosis MS or a generalized polyneuropathy (PN). A secondary endpoint for the MS arm will include spasticity and for the PN arm will be the physical examination findings of sensory changes and weakness. Meditation classes of 90 minutes duration will be led by a Buddhist monk with over 20 years experience in meditation. Sessions will be held once weekly over a 3-month period. There will be an initial introduction session that will last approximately 180 minutes for the adminsitration of formal instructions and a training session on how to do the meditation. Outcome assessments will be answered electronically on a secure system or in written form that will be able to be completed at home or at the site of the meditation class. The data will be directly downloaded into a queriable database. Outcome assessments will be based on the Short Form (SF)-36 health survey and Visual Analog Scale (VAS) for pain at baseline and at 3 months. Additionally, the Neuropathy Impairment Score (NIS) will be used for the PN pts. The PDDS spasticity questionnaire and the fatigue portion of the MSQLI for fatigue will be used for the MS patients. We plan to recruit adult patients with either MS or PN through the current patient population in the Mellen Center and Neuromuscular Center and flyers placed throughout the Cleveland Clinic. Patients will be excluded if they have performed meditation within the last 6 months, are cognitively impaired, or have an underlying illness that would preclude comprehension of the instructions. Other exclusion criteria include a history of symptomatic cardiopulmonary disease, uncontrolled HTN, current alcohol or drug abuse, and kidney or renal failure. Patients must be ambulatory and able to toilet themselves.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis OR peripheral neuropathy

Exclusion Criteria:

* Unable to walk without the assistance of others
* Unable to toilet independently
* Currently abusing drugs or alcohol
* Have performed meditation within the last 6 months
* Cognitive impairment or an underlying illness which would prevent the comprehension of instructions
* History of symptomatic/unstable heart or lung disease
* Uncontrolled high blood pressure
* Kidney or renal failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Does meditation have a beneficial effect on pain, fatigue and physical functioning in patients with multiple sclerosis and peripheral neuropathy | 2 months

SECONDARY OUTCOMES:
Does meditation lead to improvements in the neurological evaluation with regards to weakness and sensory changes with meditation. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Jinny Tavee, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No